CLINICAL TRIAL: NCT04534777
Title: Multimodal Neuroprognostication in Disorders of Consciousness
Acronym: M-Neuro-DoC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 200194
Record Dates: First submitted 2020-03-27; First posted 2020-09-01 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Consciousness Disorder
Keywords: electroencephalography; evoked potentials; functional magnetic resonance imaging; minimally conscious state; positron emission tomography; resting state fMRI (functional magnetic resonance imaging ); transcranial magnetic stimulation; traumatic brain injury; unresponsive wakefulness syndrome; vegetative state; polysomnography
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic | interventions — Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consciousness disorder patients: The overall outcome of this project will allow to draw better single-patient predictions of state, prognosis, and rehabilitation strategies and furthermore, a better understanding the pathophysiological mechanisms behind DoC that could result in groundbreaking new personalized therapeutic approaches.
  Based on the collected data, we will evaluate the respective diagnostic accuracy of all the markers acquired in clinical practice regarding the clinical outcome at 2 years.
  Interventions: Other: repeated neurological, behavioral assessments and conventional, quantitative and functional brain imagery

INTERVENTIONS:
Other: repeated neurological, behavioral assessments and conventional, quantitative and functional brain imagery — Based on the collected data, we will evaluate the respective diagnostic accuracy of all the markers acquired in clinical practice regarding the clinical outcome at 2 years.

SUMMARY:
Disorders of consciousness frequently occur at the acute phase of brain injuries. For the most severe cases, consciousness impairment can be prolonged. To optimize the medical plan and the goal of care, it is fundamental to have precise tools to predict chances of recovery of consciousness and potential disability. Currently, multimodal assessment including behavioral, neurophysiological and neuroimaging technics is recommended. However, the respective predictive values of these markers are poorly understood and decision making is challenging when results are contradictory

DETAILED DESCRIPTION:
Improved treatment of critically ill patients has resulted in increased patients' survival rates in Intensive Care Units (ICU). This is particularly true for brain injury such as traumatic brain injuries, cerebral hemorrhages or cardiac arrest. While some of these patients regain consciousness after a transient state known as coma, other will develop a prolonged disorder of consciousness (DoC) such as chronic unresponsive wakefulness syndrome (also known as vegetative state) or minimally conscious state, or will remain severely disabled. Consciousness diagnosis and prediction of recovery in DoC currently relies on standardized behavioral assessment and disease-specific markers. However, this strategy may fail to detect covert consciousness due to major sensory and motor deficits. Moreover, the DoC etiology and pathophysiology are heterogenous and most likely result from the combination of factors whose interplay still needs to be clarified. Consciousness detection in DoC is of great importance in term of medical management (e.g., pain management, communication), prognosis (e.g., orientation to adapted rehabilitation center to maximize chance of recovery) and end-of-life discussions (e.g., withholding and/or withdrawing of life support discussion). Furthermore, taking care of these patients can be very stressful due to the high levels of uncertainty associated to their potential of recovery. For all these reasons it is critical to develop personalized diagnosis and prognosis assessment tools that can allow better decisions.

The M-NeuroDoC study will take advantage from the state-of-the-art multimodal assessment ongoing at our institution for both acute and chronic patients in order to improve recovery prediction.

Indeed, our multimodal assessment practice constitutes a great and unique opportunity to better understand the respective diagnostic and prognostic accuracy performances of markers such as behavioral, electrophysiological and neuroimaging that are routinely performed at our institution.

The overall outcome of this project will allow to draw better single-patient predictions of state, prognosis, and rehabilitation strategies and furthermore, a better understanding the pathophysiological mechanisms behind DoC that could result in groundbreaking new personalized therapeutic approaches.

Based on the collected data, we will evaluate the respective diagnostic accuracy of all the markers acquired in clinical practice regarding the clinical outcome at 2 years.

Data of interest will be:

* repeated neurological assessments
* repeated behavioural assessments suing validated tools:
* neurophysiological explorations
* conventional brain imagery (CT, IRM)
* quantitative brain imagery
* functional brain imagery , mental imagery

ELIGIBILITY:
Inclusion Criteria:

1. Consciousness disorder (acute sub-acute or chronic for which our expertise is requested to better characterize the diagnostic and prognosis of recovery)
2. Brain injuries on CT or MRI (e.g. TBI) (traumatic brain-injured ), anoxia or stroke related lesions, etc…)
3. Age between 18 and 80 years

Exclusion Criteria:

1. Deep sedation (e.g. elevated ICP(intracranial pressure ), refractory status epilepticus)
2. Sever known neurodegenerative disease (e.g. Alzheimer disease)
3. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with consciousness disorder (acute sub-acute or chronic for which our expertise is requested to better characterize the diagnostic and prognosis of recovery) or with Brain injuries on CT or MRI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
prognosis accuracy of respective predictive markers of consciousness recovery | 24 MONTHS
  Calculation of the value (Chi2 tests, specificity, sensitivity, positive and negative predictive values of each tests and of their combinations to distinguish patients states and outcome (24-month GOS-E ≥ 4 or < 4).

SECONDARY OUTCOMES:
GOS-E Glasgow outcome scale - Extended | 6, 12 and 18 months
  Evolution of GOS-E (Glasgow outcome scale - Extended) scale from category 1 ==> Death to category 8: good recovery upper ==>no current problems related to the brain injury that affect daily life

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Background] Giacino JT, Kalmar K. Diagnostic and prognostic guidelines for the vegetative and minimally conscious states. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):166-74. doi: 10.1080/09602010443000498. PMID 16350959
- [Background] Hermann B, Goudard G, Courcoux K, Valente M, Labat S, Despois L, Bourmaleau J, Richard-Gilis L, Faugeras F, Demeret S, Sitt JD, Naccache L, Rohaut B; Pitie-Salpetriere hospital Neuro-ICU. Wisdom of the caregivers: pooling individual subjective reports to diagnose states of consciousness in brain-injured patients, a monocentric prospective study. BMJ Open. 2019 Feb 21;9(2):e026211. doi: 10.1136/bmjopen-2018-026211. PMID 30792234
- [Background] Andre-Obadia N, Zyss J, Gavaret M, Lefaucheur JP, Azabou E, Boulogne S, Guerit JM, McGonigal A, Merle P, Mutschler V, Naccache L, Sabourdy C, Trebuchon A, Tyvaert L, Vercueil L, Rohaut B, Delval A. Recommendations for the use of electroencephalography and evoked potentials in comatose patients. Neurophysiol Clin. 2018 Jun;48(3):143-169. doi: 10.1016/j.neucli.2018.05.038. Epub 2018 May 18. PMID 29784540
- [Background] Balanca B, Dailler F, Boulogne S, Ritzenthaler T, Gobert F, Rheims S, Andre-Obadia N. Diagnostic accuracy of quantitative EEG to detect delayed cerebral ischemia after subarachnoid hemorrhage: A preliminary study. Clin Neurophysiol. 2018 Sep;129(9):1926-1936. doi: 10.1016/j.clinph.2018.06.013. Epub 2018 Jul 5. PMID 30007892
- [Derived] Rohaut B, Calligaris C, Hermann B, Perez P, Faugeras F, Raimondo F, King JR, Engemann D, Marois C, Le Guennec L, Di Meglio L, Sangare A, Munoz Musat E, Valente M, Ben Salah A, Demertzi A, Belloli L, Manasova D, Jodaitis L, Habert MO, Lambrecq V, Pyatigorskaya N, Galanaud D, Puybasset L, Weiss N, Demeret S, Lejeune FX, Sitt JD, Naccache L. Multimodal assessment improves neuroprognosis performance in clinically unresponsive critical-care patients with brain injury. Nat Med. 2024 Aug;30(8):2349-2355. doi: 10.1038/s41591-024-03019-1. Epub 2024 May 30. PMID 38816609